CLINICAL TRIAL: NCT00638690
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Abiraterone Acetate (CB7630) Plus Prednisone in Patients With Metastatic Castration-Resistant Prostate Cancer Who Have Failed Docetaxel-Based Chemotherapy
Brief Title: Abiraterone Acetate in Castration-Resistant Prostate Cancer Previously Treated With Docetaxel-Based Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016924; COU-AA-301 (Other: Cougar Biotechnology, Inc)
Record Dates: First submitted 2008-03-13; First posted 2008-03-19 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Prostatic Neoplasms
Keywords: Metastatic Castration-Resistant Prostate Cancer; CRPC; Abiraterone Acetate; CB7630
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abiraterone acetate plus prednisone/prednisolone (Experimental)
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone/prednisolone
- Placebo plus prednisone/prednisolone (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Prednisone/prednisolone

INTERVENTIONS:
Drug: Placebo — Four tablets once daily until disease progression
  Arms: Placebo plus prednisone/prednisolone
Drug: Abiraterone acetate — Four 250-mg tablets once daily until disease progression
  Arms: Abiraterone acetate plus prednisone/prednisolone
Drug: Prednisone/prednisolone — 5 mg twice daily until disease progression

SUMMARY:
This is a phase 3 study to compare the clinical benefit of abiraterone acetate plus prednisone with placebo plus prednisone in patients with metastatic castration-resistant prostate cancer (CRPC) who have failed one or two chemotherapy regimens. At least one of the previous chemotherapies must have contained docetaxel.

DETAILED DESCRIPTION:
Abiraterone acetate is a steroidal irreversible inhibitor of CYP17 (17α hydroxylase/C17, 20-lyase), blocking 2 important enzymatic activities in the synthesis of testosterone. The goal of this study is to compare the clinical benefit of abiraterone acetate plus prednisone with placebo plus prednisone in patients with metastatic castration-resistant prostate cancer (CRPC) who have failed one or two chemotherapy regimens, one of which contains docetaxel. All patients involved in the study will be randomized (assigned by chance) into one of two arms and will not know what study drug is being given to them. Study drug randomization allocation will be 2:1 (abiraterone acetate: placebo). The study will be conducted in the United States, Canada, Australia, and the EU. The study will consist of screening, treatment, and follow-up. In this study, patients will receive study treatment (abiraterone acetate or placebo) plus prednisone until progression of clinical disease. Follow-up will continue until patient dies, is lost to follow-up, or withdraws informed consent. After providing written informed consent, patients will have screening procedures completed to determine eligibility. Safety evaluations at the screening procedure will include a physical examination, vital signs, and clinical blood laboratory tests, ECG, radiographs, urine tests, and recording of any adverse events including details of current prostate cancer symptoms. Patients will be asked to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 13 weeks after last study drug administration.

Study medication, abiraterone acetate,is an oral (by mouth) medication to be administered as four (4) 250mg abiraterone acetate tablets or 4 placebo tablets to be taken at least one hour before or two hours after a meal anytime up to 10PM everyday. Prednisone will be administered as 5mg orally twice a day for both groups. Each cycle will be 28 days. Study treatment will continue until disease progression as determined by investigator or when the patient meets criteria for withdrawal from study.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Castration-Resistant Prostate Cancer Progression after one or two prior cytotoxic chemotherapies
* At least one chemotherapy must have contained docetaxel
* Eastern Cooperative Oncology Group (ECOG) Performance Status <= 2
* Medical or surgical castration with testosterone < 50 ng/dL
* Adequate bone marrow, hepatic and renal function
* Potassium >= 3.5 mmol/L
* Able to swallow the study drug whole as a tablet
* Informed Consent

Exclusion Criteria:

* More than two prior cytotoxic chemotherapy regimens
* Prior Ketoconazole for prostate cancer
* Prior abiraterone acetate or other CYP17 inhibitor or investigational agents targeting the androgen receptor for prostate cancer
* Uncontrolled hypertension
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease
* Other malignancy
* Known brain metastasis
* GI disorder affecting absorption
* Not willing to use contraception

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1195 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (127):
- United States (54):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Beverly Hills, California
  - Duarte, California
  - Los Angeles, California
  - Marina del Rey, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Bristol, Connecticut
  - New Haven, Connecticut
  - Stamford, Connecticut
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Galesburg, Illinois
  - Indianapolis, Indiana
  - Westwood, Kansas
  - Wichita, Kansas
  - Marrero, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Robbinsdale, Minnesota
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Box 302, New York
  - East Setauket, New York
  - New Hyde Park, New York
  - New York, New York
  - Stony Brook, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Myrtle Beach, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Virgiania Beach, Virginia
  - Seattle, Washington
- Australia (17):
  - Adelaide
  - Camperdown
  - Footscray
  - Geelong
  - Heidelberg
  - Herston
  - Hobart
  - Hornsby
  - Kogarah
  - Kurralta Park
  - Liverpool
  - Milton
  - Parkville
  - Perth
  - Subiaco
  - Wodonga
  - Wollongong
- Austria (3):
  - Linz
  - Salzburg
  - Vienna
- Belgium (9):
  - Antwerp
  - Bonheiden
  - Brussels
  - Ghent
  - Hasselt
  - Kortrijk
  - Leuven
  - Liège
  - Roeselare
- Canada (11):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Regina, Saskatchewan
  - Calgary Ab
  - London
- France (9):
  - Angers
  - Caen
  - Cannes
  - Dijon
  - Lyon
  - Paris
  - Saint-Herblain
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (5):
  - Aachen
  - Berlin
  - Dresden
  - Hamburg
  - Homburg/Saar
- Hungary (2):
  - Pécs
  - Szombathely
- Ireland (2):
  - Cork
  - Dublin
- Nijmegen, Netherlands
- Spain (3):
  - Badalona
  - Barcelona
  - Madrid
- United Kingdom (11):
  - Belfast
  - Birmingham
  - Cambridge
  - Glasgow
  - London
  - Manchester
  - Newcastle upon Tyne
  - Northwood
  - Oxford
  - Sutton
  - Whitchurch

REFERENCES:
- [Derived] Heller G, McCormack R, Kheoh T, Molina A, Smith MR, Dreicer R, Saad F, de Wit R, Aftab DT, Hirmand M, Limon A, Fizazi K, Fleisher M, de Bono JS, Scher HI. Circulating Tumor Cell Number as a Response Measure of Prolonged Survival for Metastatic Castration-Resistant Prostate Cancer: A Comparison With Prostate-Specific Antigen Across Five Randomized Phase III Clinical Trials. J Clin Oncol. 2018 Feb 20;36(6):572-580. doi: 10.1200/JCO.2017.75.2998. Epub 2017 Dec 22. PMID 29272162
- [Derived] Chi KN, Kheoh T, Ryan CJ, Molina A, Bellmunt J, Vogelzang NJ, Rathkopf DE, Fizazi K, Kantoff PW, Li J, Azad AA, Eigl BJ, Heng DY, Joshua AM, de Bono JS, Scher HI. A prognostic index model for predicting overall survival in patients with metastatic castration-resistant prostate cancer treated with abiraterone acetate after docetaxel. Ann Oncol. 2016 Mar;27(3):454-60. doi: 10.1093/annonc/mdv594. Epub 2015 Dec 18. PMID 26685010
- [Derived] Fizazi K, Flaig TW, Stockle M, Scher HI, de Bono JS, Rathkopf DE, Ryan CJ, Kheoh T, Li J, Todd MB, Griffin TW, Molina A, Ohlmann CH. Does Gleason score at initial diagnosis predict efficacy of abiraterone acetate therapy in patients with metastatic castration-resistant prostate cancer? An analysis of abiraterone acetate phase III trials. Ann Oncol. 2016 Apr;27(4):699-705. doi: 10.1093/annonc/mdv545. Epub 2015 Nov 25. PMID 26609008
- [Derived] Antoun S, Bayar A, Ileana E, Laplanche A, Fizazi K, di Palma M, Escudier B, Albiges L, Massard C, Loriot Y. High subcutaneous adipose tissue predicts the prognosis in metastatic castration-resistant prostate cancer patients in post chemotherapy setting. Eur J Cancer. 2015 Nov;51(17):2570-7. doi: 10.1016/j.ejca.2015.07.042. Epub 2015 Aug 13. PMID 26278649
- [Derived] Xu XS, Ryan CJ, Stuyckens K, Smith MR, Saad F, Griffin TW, Park YC, Yu MK, Vermeulen A, Poggesi I, Nandy P. Correlation between Prostate-Specific Antigen Kinetics and Overall Survival in Abiraterone Acetate-Treated Castration-Resistant Prostate Cancer Patients. Clin Cancer Res. 2015 Jul 15;21(14):3170-7. doi: 10.1158/1078-0432.CCR-14-1549. Epub 2015 Mar 31. PMID 25829400
- [Derived] Scher HI, Heller G, Molina A, Attard G, Danila DC, Jia X, Peng W, Sandhu SK, Olmos D, Riisnaes R, McCormack R, Burzykowski T, Kheoh T, Fleisher M, Buyse M, de Bono JS. Circulating tumor cell biomarker panel as an individual-level surrogate for survival in metastatic castration-resistant prostate cancer. J Clin Oncol. 2015 Apr 20;33(12):1348-55. doi: 10.1200/JCO.2014.55.3487. Epub 2015 Mar 23. PMID 25800753
- [Derived] Mulders PF, Molina A, Marberger M, Saad F, Higano CS, Chi KN, Li J, Kheoh T, Haqq CM, Fizazi K. Efficacy and safety of abiraterone acetate in an elderly patient subgroup (aged 75 and older) with metastatic castration-resistant prostate cancer after docetaxel-based chemotherapy. Eur Urol. 2014 May;65(5):875-83. doi: 10.1016/j.eururo.2013.09.005. Epub 2013 Sep 20. PMID 24099659
- [Derived] Harland S, Staffurth J, Molina A, Hao Y, Gagnon DD, Sternberg CN, Cella D, Fizazi K, Logothetis CJ, Kheoh T, Haqq CM, de Bono JS, Scher HI; COU-AA-301 Investigators. Effect of abiraterone acetate treatment on the quality of life of patients with metastatic castration-resistant prostate cancer after failure of docetaxel chemotherapy. Eur J Cancer. 2013 Nov;49(17):3648-57. doi: 10.1016/j.ejca.2013.07.144. Epub 2013 Aug 22. PMID 23973186
- [Derived] Ryan CJ, Molina A, Li J, Kheoh T, Small EJ, Haqq CM, Grant RP, de Bono JS, Scher HI. Serum androgens as prognostic biomarkers in castration-resistant prostate cancer: results from an analysis of a randomized phase III trial. J Clin Oncol. 2013 Aug 1;31(22):2791-8. doi: 10.1200/JCO.2012.45.4595. Epub 2013 Jul 1. PMID 23816964
- [Derived] Logothetis CJ, Basch E, Molina A, Fizazi K, North SA, Chi KN, Jones RJ, Goodman OB, Mainwaring PN, Sternberg CN, Efstathiou E, Gagnon DD, Rothman M, Hao Y, Liu CS, Kheoh TS, Haqq CM, Scher HI, de Bono JS. Effect of abiraterone acetate and prednisone compared with placebo and prednisone on pain control and skeletal-related events in patients with metastatic castration-resistant prostate cancer: exploratory analysis of data from the COU-AA-301 randomised trial. Lancet Oncol. 2012 Dec;13(12):1210-7. doi: 10.1016/S1470-2045(12)70473-4. Epub 2012 Nov 9. PMID 23142059
- [Derived] Fizazi K, Scher HI, Molina A, Logothetis CJ, Chi KN, Jones RJ, Staffurth JN, North S, Vogelzang NJ, Saad F, Mainwaring P, Harland S, Goodman OB Jr, Sternberg CN, Li JH, Kheoh T, Haqq CM, de Bono JS; COU-AA-301 Investigators. Abiraterone acetate for treatment of metastatic castration-resistant prostate cancer: final overall survival analysis of the COU-AA-301 randomised, double-blind, placebo-controlled phase 3 study. Lancet Oncol. 2012 Oct;13(10):983-92. doi: 10.1016/S1470-2045(12)70379-0. Epub 2012 Sep 18. PMID 22995653
- [Derived] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate: Abiraterone acetate plus prednisone/prednisolone administered as four 250 mg tablets of abiraterone acetate once daily plus 5 mg prednisone/5 mg prednisolone twice daily until disease progression.
- Placebo: Placebo plus prednisone/prednisolone administered as four placebo tablets once daily plus 5 mg prednisone/5 mg prednisolone tablet twice daily until disease progression.
Period: Overall Study
Arm/Group | Abiraterone Acetate | Placebo
Started | 797 | 398
Completed | 116 | 56
Not Completed | 681 | 342
Not completed — Death | 655 | 335
Not completed — Withdrawal by Subject | 22 | 5
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo plus prednisone/prednisolone
- Total: Total of all reporting groups
Arm/Group | Abiraterone Acetate | Placebo | Total
Number analyzed (Participants) | 797 | 398 | 1195
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.4) | 68.9 (8.61) | 69 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 797 | 398 | 1195
Region of Enrollment [Number; unit: participants]
  Australia | 69 | 35 | 104
  Austria | 11 | 1 | 12
  Belgium | 32 | 11 | 43
  Canada | 97 | 57 | 154
  France | 57 | 33 | 90
  Germany | 26 | 12 | 38
  Hungary | 5 | 2 | 7
  Italy | 21 | 12 | 33
  Netherlands | 4 | 2 | 6
  Republic of Ireland | 7 | 7 | 14
  Spain | 13 | 3 | 16
  United Kingdom | 119 | 61 | 180
  United States | 336 | 162 | 498

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time interval from the date of randomization to the date of death from any cause.
Time Frame: Up to 60 months
Population: Analysis was performed on the Intent-to-Treat (ITT) population. The ITT population is composed of all patients randomized into the study and who will be classified according to their assigned teatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abiraterone Acetate | Placebo
Number analyzed (Participants) | 797 | 398
Days | 450.0 [430.0 to 470.0] | 332.0 [310.0 to 366.0]
Statistical Analysis 1: Comparison: Abiraterone Acetate vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Nominal P-value is 0.0142 at interim analysis based on group sequential design; This was a stratified analysis; Hazard Ratio (HR) = 0.646, 95% CI 2-sided [0.543 to 0.768]

2. Secondary Outcome: Time to Prostate-Specific Antigen Progression According to Prostate Specific Antigen Working Group Criteria
Description: The time interval from the date of randomization to the date of the prostate-specific antigen (PSA) progression as defined in the protocol-specific Prostate Specific Antigen Working Group (PSAWG) criteria, namely, a PSA level of at least 5 ng/ml that has risen on at least 2 successive occasions, at least 2 weeks apart.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abiraterone Acetate | Placebo
Number analyzed (Participants) | 797 | 398
Days | 309.0 [255.0 to 421.0] | 200.0 [170.0 to 254.0]
Statistical Analysis 1: Comparison: Abiraterone Acetate vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Nominal P-value = 0.05; This was a stratified analysis; Hazard Ratio (HR) = 0.580, 95% CI [0.462 to 0.728]

3. Secondary Outcome: Number of Patients Achieving a Prostate-Specific Antigen Decline >=50%
Description: A prostate-specific antigen (PSA) response was defined as a >=50% decline from baseline.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Abiraterone Acetate | Placebo
Number analyzed (Participants) | 797 | 398
Participants | 232 | 22
Statistical Analysis 1: Comparison: Abiraterone Acetate vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared — Nominal P-value = 0.05; Risk Ratio (RR) = 5.266, 95% CI 2-sided [3.459 to 8.018]

4. Secondary Outcome: Radiographic Progression-free Survival
Description: Radiographic progression-free survival is based on imaging studies according to modified Response Evaluation Criteria in Solid Tumors (RECIST): baseline lymph node size must be >=2.0 cm to be considered a target lesion; progression on bone scans with >=2 new lesions not consistent with tumor flare, confirmed on a second scan >=6 weeks later that shows >=1 additional new lesion.
Time Frame: Up to 11 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abiraterone Acetate | Placebo
Number analyzed (Participants) | 797 | 398
Days | 171.0 [169.0 to 192.0] | 110.0 [88.0 to 168.0]
Statistical Analysis 1: Comparison: Abiraterone Acetate vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — The nominal P-value = 0.05; This was a stratified analysis; Hazard Ratio (HR) = 0.673, 95% CI 2-sided [0.585 to 0.776]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Following interim analysis of the study by the Independent Data Monitoring Committee in August 2010, the protocol was amended to provide for the unblinding of all study participants and the option for placebo participants to receive abiraterone acetate treatment; 67 placebo participants crossed over.
Groups:
- Placebo to Abiraterone Acetate: Placebo plus prednisone/prednisolone crossed over to abiraterone acetate plus prednisone/prednisolone
Arm/Group | Abiraterone Acetate | Placebo | Placebo to Abiraterone Acetate
Serious Adverse Events (participants affected / at risk) | 365/791 | 175/394 | 29/67
Other Adverse Events (participants affected / at risk) | 766/791 | 381/394 | 57/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=791) | Placebo (N=394) | Placebo to Abiraterone Acetate (N=67)
Anaemia (Blood and lymphatic system disorders) | 26 | 15 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperglycaemia (Endocrine disorders) | 0 | 1 | 0
Blindness (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 3 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 17 | 9 | 1
Malaise (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 6 | 0
Pyrexia (General disorders) | 6 | 9 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 21 | 5 | 3
Pyelonephritis (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 14 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 4 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 14 | 4 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Convulsion (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Epiduritis (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Hemiparesis (Nervous system disorders) | 2 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 3 | 2 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 12 | 11 | 0
Hydronephrosis (Renal and urinary disorders) | 12 | 3 | 2
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0
Hypotension (Vascular disorders) | 4 | 1 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 3 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 3 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 7 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0 | 0
Adrenal suppression (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Pupils unequal (Eye disorders) | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 9 | 1 | 0
Catheter related complication (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 12 | 2 | 2
Fatigue (General disorders) | 9 | 6 | 1
General physical health deterioration (General disorders) | 5 | 2 | 0
Generalised oedema (General disorders) | 2 | 0 | 0
Hernia obstructive (General disorders) | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 0
Oedema peripheral (General disorders) | 3 | 0 | 0
Performance status decreased (General disorders) | 1 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 2 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Candida sepsis (Infections and infestations) | 0 | 1 | 0
Catheter sepsis (Infections and infestations) | 1 | 0 | 0
Central line infection (Infections and infestations) | 2 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Genitourinary tract infection (Infections and infestations) | 0 | 1 | 0
Groin infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Kidney infection (Infections and infestations) | 2 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 3 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Lung infection (Infections and infestations) | 3 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia escherichia (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Staphylococcal infection (Infections and infestations) | 3 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 19 | 3 | 3
Wound infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 5 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pathological fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 3 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 11 | 4
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 16 | 13 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 7 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Brachial plexopathy (Nervous system disorders) | 0 | 1 | 0
Brain compression (Nervous system disorders) | 0 | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Bulbar palsy (Nervous system disorders) | 0 | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 0 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0 | 0
Cranial neuropathy (Nervous system disorders) | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 1 | 0
Nerve root lesion (Nervous system disorders) | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 23 | 18 | 3
Subdural hygroma (Nervous system disorders) | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 2 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 4 | 3 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Bladder stenosis (Renal and urinary disorders) | 0 | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 3 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 4 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 7 | 5 | 2
Renal impairment (Renal and urinary disorders) | 3 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 3 | 1 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 9 | 6 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Eye muscle recession (Surgical and medical procedures) | 0 | 1 | 0
Malignant tumour excision (Surgical and medical procedures) | 1 | 0 | 0
Pain management (Surgical and medical procedures) | 1 | 0 | 0
Ureteral stent insertion (Surgical and medical procedures) | 0 | 1 | 0
Cardiovascular insufficiency (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Superior vena caval occlusion (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=791) | Placebo (N=394) | Placebo to Abiraterone Acetate (N=67)
Anaemia (Blood and lymphatic system disorders) | 202 | 105 | 11
Constipation (Gastrointestinal disorders) | 236 | 124 | 14
Diarrhoea (Gastrointestinal disorders) | 166 | 57 | 13
Dyspepsia (Gastrointestinal disorders) | 54 | 15 | 4
Nausea (Gastrointestinal disorders) | 272 | 132 | 19
Vomiting (Gastrointestinal disorders) | 204 | 97 | 14
Pyrexia (General disorders) | 87 | 28 | 7
Nasopharyngitis (Infections and infestations) | 58 | 25 | 6
Contusion (Injury, poisoning and procedural complications) | 70 | 22 | 3
Anorexia (Metabolism and nutrition disorders) | 155 | 74 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 61 | 20 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 149 | 36 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 246 | 93 | 20
Dizziness (Nervous system disorders) | 99 | 40 | 2
Headache (Nervous system disorders) | 111 | 42 | 6
Anxiety (Psychiatric disorders) | 55 | 21 | 2
Depression (Psychiatric disorders) | 47 | 21 | 2
Insomnia (Psychiatric disorders) | 98 | 52 | 5
Haematuria (Renal and urinary disorders) | 76 | 27 | 2
Nocturia (Renal and urinary disorders) | 54 | 17 | 4
Pollakiuria (Renal and urinary disorders) | 61 | 21 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 116 | 33 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 117 | 49 | 10
Hypertension (Vascular disorders) | 79 | 27 | 5
Abdominal pain (Gastrointestinal disorders) | 111 | 45 | 4
Dry mouth (Gastrointestinal disorders) | 61 | 20 | 4
Asthenia (General disorders) | 131 | 54 | 5
Fatigue (General disorders) | 384 | 172 | 19
Oedema peripheral (General disorders) | 228 | 75 | 11
Pain (General disorders) | 40 | 15 | 2
Upper respiratory tract infection (Infections and infestations) | 57 | 11 | 2
Urinary tract infection (Infections and infestations) | 100 | 27 | 6
Weight decreased (Investigations) | 110 | 57 | 4
Decreased appetite (Metabolism and nutrition disorders) | 89 | 36 | 4
Dehydration (Metabolism and nutrition disorders) | 43 | 18 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 282 | 138 | 23
Bone pain (Musculoskeletal and connective tissue disorders) | 219 | 112 | 12
Groin pain (Musculoskeletal and connective tissue disorders) | 51 | 22 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 79 | 37 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 94 | 38 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 140 | 56 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 50 | 17 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 35 | 20 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 170 | 81 | 13
Hypoaesthesia (Nervous system disorders) | 41 | 15 | 2
Paraesthesia (Nervous system disorders) | 41 | 15 | 3
Urinary incontinence (Renal and urinary disorders) | 42 | 15 | 4
Pelvic pain (Reproductive system and breast disorders) | 20 | 20 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 17 | 12 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 44 | 16 | 1
Hot flush (Vascular disorders) | 157 | 68 | 2
Hypotension (Vascular disorders) | 35 | 18 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 60 days from the time submitted to the sponsor for review. After 1) publication of multi-center results, 2) notification by sponsor that a multi-center submission is no longer planned, or 3) the 18 month anniversary of the termination of the study at all sites, the institution and investigator may publish or publicly present study data.